CLINICAL TRIAL: NCT04247594
Title: A Phase 2, Open Label, Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Voxelotor in Patients With Sickle Cell Disease
Brief Title: Dose Escalation Study to Evaluate the Safety, Tolerability, PK and PD of Voxelotor in Patients With SCD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data will not inform further development of Voxelotor
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-029; C5341042 (Other: Alias Study Number)
Record Dates: First submitted 2020-01-21; First posted 2020-01-30 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease, SCD
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Period 1 (Experimental): 1500 mg per day
  Interventions: Drug: Voxelotor
- Period 2 (Experimental): 2000 mg per day
  Interventions: Drug: Voxelotor
- Period 3 (Experimental): 2500 mg per day
  Interventions: Drug: Voxelotor
- Period 4 (Experimental): 3000 mg per day
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — synthetic small molecule supplied as 500 mg tablets

SUMMARY:
Study participants will undergo up to four periods of voxelotor administered orally at progressively higher dose levels from 1500 mg until either a maximum tolerated dose (MTD) or 3000 mg/day dose is reached, whichever occurs first

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with SCD
2. Documentation of SCD genotype HbSS or HbSB0
3. Age 18 to < 60 years, inclusive
4. Hemoglobin ≥ 5.5 and ≤ 10.5 g/dL during Screening, and considered stable and close to Baseline by the Investigator
5. For participants taking HU, the dose in mg/kg must be stable for at least 90 days prior to signing the informed consent form (ICF) and with no anticipated need for dose adjustments during the study, in the opinion of the Investigator.
6. Participants, who if female and of child-bearing potential, agree to use highly effective methods of contraception or practicing abstinence from study start to 30 days after the last dose of study drug, and who if male, agree to use barrier methods of contraception or practice abstinence from study start to 30 days after the last dose of study drug
7. Participant has provided documented informed consent

Exclusion Criteria:

1. More than 10 VOCs within 12 months of screening that required a hospital, emergency room, or clinic visit
2. Female participant who is breast feeding or pregnant
3. Receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion) or have received an RBC transfusion for any reason within 60 days of signing the ICF or at any time during the Screening Period
4. Hospitalized for sickle cell crisis or other vaso-occlusive event within 30 days prior to dosing (ie, a vaso-occlusive event cannot be within 30 days prior to dosing)
5. Screening laboratory test of alanine aminotransferase (ALT) > 4 × upper level of normal (ULN)
6. Clinically significant bacterial, fungal, parasitic, or viral infection which requires therapy, including acute bacterial infection requiring antibiotics
7. Known to be COVID-19 positive from within 3 weeks of screening through Day 1
8. Participants with active hepatitis A, B, or C or who are known to be human immunodeficiency virus (HIV) positive
9. Severe renal dysfunction (estimated glomerular filtration rate < 30 mL/min/1.73 m2 at the Screening visit; calculated by the local laboratory to assess safety) or is on chronic dialysis
10. History of malignancy within the past 2 years prior to treatment Day 1 requiring chemotherapy and/or radiation (with the exception of local therapy for non-melanoma skin malignancy)
11. History of unstable or deteriorating cardiac or pulmonary disease within 6 months prior to consent including but not limited to the following:

    1. Unstable angina pectoris or myocardial infarction or elective coronary intervention
    2. Congestive heart failure requiring hospitalization
    3. Uncontrolled clinically significant arrhythmias
    4. Pulmonary hypertension
12. Criteria related to ECG parameters:

    1. PR interval > 220 msec in any participant
    2. QRS interval > 120 msec or QT interval corrected using Fridericia's formula (QTcF) > 480 msec (both genders) in participants without bundle branch block
    3. QRS interval > 120 msec in participants with newly (within 3 months) emerged bundle branch block
    4. A participant with stable bundle branch block with or without stable cardiac disease may be enrolled; QRS interval > 120 msec and QTcF interval > 480 msec are acceptable in these participants.
13. Any condition affecting drug absorption, such as major surgery involving the stomach or small intestine (prior cholecystectomy is acceptable)
14. Participated in another clinical trial of an investigational agent or medical device within 30 days or 5 half-lives of date of informed consent, whichever is longer, or is currently participating in another trial of an investigational agent or medical device
15. Inadequate venous access as determined by the Investigator/site staff
16. Medical, psychological, or behavioral conditions, which, in the opinion of the Investigator, may preclude safe participation, confound study interpretation, interfere with compliance, or preclude informed consent
17. Received erythropoietin or other hematopoietic growth factor treatment within 28 days of signing ICF or is anticipated to require such agents during the study
18. Ongoing or recent (within 2 years) substance abuse
19. Known allergy to voxelotor
20. Use of herbal medications (eg, St. John's Wort), sensitive cytochrome P450 (CYP) 3A4 substrates with a narrow therapeutic index, strong CYP3A4 inhibitors, fluconazole, or moderate or strong CYP3A4 inducers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United Kingdom (6):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Guy's Hospital, London
  - Hammersmith Hospital, London
  - Homerton University, London
  - King's College Hospital, London
  - Royal London Hospital, Barts Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each individual was provided with oral and written information describing the nature, purpose and duration of the study, participation/termination conditions, and risks and benefits. Prior to initiation of any study-related procedures, subjects signed and dated the ICF to participate in the study.
Pre-assignment Details: All patients completed the following study procedures prior to a confirmation of eligibility: Signed Informed Consent Form, Review inclusion/exclusion criteria, Medication and Medical History, Height/Weight/ BMI, Vital signs, ECG (12-lead) in triplicate, Physical examination, Serum pregnancy test (females of child-bearing potential only) and so on.
Groups:
- Open Label: Participants will receive progressively higher doses of voxelotor administration starting from 1500 mg Voxelotor: synthetic small molecule supplied as 500 mg tablets
Period: Overall Study
Arm/Group | Open Label
Started | 6
Completed | 2
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Subjects treated with at least one dose of Voxelotor
Arm/Group | Open Label
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 32 [27 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 6
Weight [Median (Full Range); unit: kg] | 66.45 [47 to 74.9]
Height [Median (Full Range); unit: cm] | 171 [163 to 190]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 22 [18 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (AEs)
Description: Treatment emergent AEs including SAEs
Time Frame: approximately 300 days
Population: Subjects treated with at least one dose of voxelotor
Measure: Count of Participants; unit: Participants
Groups:
- Voxelotor 1500 mg: Participants received 1500 mg voxelotor per day for 3 weeks in Period 1.
- Voxelotor 2000 mg: Participants received 2000 mg voxelotor per day for 3 weeks in Period 2.
- Voxelotor 2500 mg: Participants received 2500 mg voxelotor per day for 3 weeks in Period 3.
- Voxelotor 3000 mg: Participants received 3000 mg voxelotor per day for 3 weeks in Period 4.
Arm/Group | Voxelotor 1500 mg | Voxelotor 2000 mg | Voxelotor 2500 mg | Voxelotor 3000 mg
Number analyzed (Participants) | 6 | 4 | 3 | 1
Participants
  Sickle cell disease (SCD) related TEAE | 5 | 1 | 1 | 0
  Non-SCD related TEAE | 6 | 4 | 2 | 1

2. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Hb, Unconjugated Bilirubin, % Reticulocyte, Absolute Reticulocyte, and Lactate Dehydrogenase [LDH]
Time Frame: approximately 200 days
Population: Subjects treated with at least one dose of Voxelotor
Measure: Count of Participants; unit: Participants
Arm/Group | Voxelotor 1500 mg | Voxelotor 2000 mg | Voxelotor 2500 mg | Voxelotor 3000 mg
Number analyzed (Participants) | 6 | 4 | 3 | 1
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With an Hb Increase > 1 g/dL Compared to Baseline
Description: Participants with an Hb increase > 1 g/dL compared to Baseline.
Time Frame: approximately 200 days
Population: Subjects treated with at least one dose of Voxelotor
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Incidence Rate of VOCs
Description: Incidence rate of vaso-occlusive crisis
Time Frame: approximately 200 days
Population: Subjects treated with at least one dose of Voxelotor
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: All adverse events were recorded from the time the study participant signs the informed consent form (ICF) until 28 days after the last dose of study drug (up to approximately 300 days)
Description: Adverse events were coded using the Medical Dictionary for Regulatory Activities Dictionary (MedDRA) version 24.0 and were categorized by system organ class (SOC) and preferred term (PT). National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 was used to determine the grade.
Arm/Group | Period 1 | Period 2 | Period 3 | Period 4
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/4 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 2/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 (N=6) | Period 2 (N=4) | Period 3 (N=3) | Period 4 (N=1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 (N=6) | Period 2 (N=4) | Period 3 (N=3) | Period 4 (N=1)
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT04247594/Prot_SAP_000.pdf